CLINICAL TRIAL: NCT01927653
Title: Imaging the Neural Network Connectivity on Patients With Mild Cognitive Impairment
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wang . Jiun-Jie, Study Principal Investigator, Chang Gung Memorial Hospital
Other Study IDs: 98-3628B
Record Dates: First submitted 2013-06-19; First posted 2013-08-22 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Mild Cognitive Impairment
Keywords: Amnestic mild cognitive impairment; Dysexecutive mild cognitive impairment; Diffusion MRI
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- The patients with amnestic MCI: The patients with single domain amnestic MCI have a Clinical Dementia Rating score of 0.5 with isolated memory impairment without deficits in other cognitive domains. A cutoff scores below 1.5 Standard Deviation (SD) (or 7 percentile) of one of the tests in domains of cognitions employed psychometric tests; They should meet the following criteria:
  1. memory complaint
  2. normal general cognition
  3. normal activities of daily living
  4. not demented
- The patients with dysexecutive MCI: The patients of dMCI have relatively focal dysfunction in executive domain with the tests of memory, language and visuospatial skills within normal limits. The patients with single domain dysexecutive MCI should meet the following criteria:
  1. relatively focal executive dysfunction
  2. Within reference range on tests of memory, language and visuospatial skills
  3. normal general cognition
  4. normal activities of daily living
  5. not demented
- The healthy volunteers: The healthy volunteers should be normal neuropsychological assessments as well as CDR=0 without significant neuropsychiatric disorder, right-handed, gender balanced and meet the following criteria:
  1. Age and gender matched healthy subjects without significant neuropsychiatric disorder
  2. Able to understand and provide signed informed consent

SUMMARY:
The hypothesis tested if the diffusion properties in the base line, such as mean diffusivity or kurtosis, can differentiate two subtypes of MCI and predict the clinical outcome in Patients. The hypothesis further supports the correlation of the measured diffusion properties and the disease severity. We therefore proposed to investigate the potential value of diffusion properties as a possible tool to monitor the disease progression. The disease related changes in neural connectivity will be investigated.

1. The diffusion MRI could provide an improved diagnosis of Alzheimer's Disease and Mild cognitive Impairment.

   Explanation:

   The deposition of the macromolecules such as beta amyloid in the brain and the associated neuron death of the patient could lead to observable changes in tissue microenvironment. The related changes would lead to alterations in either the amplitude or distribution of water diffusion. In turn it could be detected in diffusion tensor and kurtosis.
2. aMCI is a preclinical state of AD and dMCI is from a different etiology, which can be differentially diagnosis by MRI. Diffusion Imaging could help to predict the clinical outcome Explanation

DETAILED DESCRIPTION:
Mild Cognitive Impairment (MCI) referred to a decline of cognition in elder adults that are not of sufficient magnitude to meet the criteria for dementia. It is usually regarded as a transition state between patients of Alzheimer's Disease (AD) and the age matched healthy adults. It is a heterogeneous syndrome which can be divided into two subtypes: amnestic and dysexecutive. This 3 year proposal continues from a NSc funded project, in which we reported that the amnestic MCI could involve global white matter changes and therefore could be a preclinical status to AD. In contrast, no compromise in white matter status was found in patients of dysexecutive MCI. Therefore we proposed to further investigate the phenomena in this project.

The subjects will be divided into 3 groups: 30 patients with amnestic MCI, 30 with dysexecutive MCI and 30 healthy age-matched normal controls. Comprehensive neuropsychological examinations will be performed after detailed clinical history and physical screening, including Mini-Mental Status Examination, Clinical Dementia Rating and the Cognitive Abilities Screening Instrument. Successful candidate will be examined by 3T MRI, including diffusion imaging and high resolution T1 weighted anatomical images.

The current project proposed to examine the sensitivity and specificity of diffusion Magnetic Resonance Imaging, in the diagnosis of MCI and differential diagnosis of two subtypes. Both the conventional tensor derived indices and diffusion kurtosis will be compared. This is due to the fact that in a recently publication in Radiology, we reported an improved diagnostic performance on neurodegenerative disease from diffusion kurtosis than diffusion tensor. Secondly we will examine the regional changes of diffusion properties and correlated with the white matter involvement in patients. High resolution track density images will be implemented and compared with the susceptibility weighted imaging in an effort to address the underlying changes in pathophysiology. In the third year, the prognostic value of diffusion MRI will be determined. The optimal cutoff value of diffusion MRI in the prediction of conversion to Alzheimer's disease will be reported. The diffusion properties in patients with early conversion (the 2nd year) and late conversion (the 3rd year) will be compared.

It is expected that changes in diffusion can be used as an image based surrogate marker during the neurodegenerative process. The new insight into the temporal evolution of the diffusion MRI might help to understand the underlying etiology and pathophysiology between the amnestic and dysexecutive MCI patients, which can contribute to an early intervention strategy and might ultimately lead to an effective treatment.

ELIGIBILITY:
Inclusion Criteria:

The patients with amnestic MCI

The patients with single domain amnestic MCI have a Clinical Dementia Rating score of 0.5 with isolated memory impairment without deficits in other cognitive domains. A cutoff scores below 1.5 Standard Deviation (SD) (or 7 percentile) of one of the tests in domains of cognitions employed psychometric tests; They should meet the following criteria:

1. memory complaint
2. normal general cognition
3. normal activities of daily living
4. not demented

The patients with dysexecutive MCI

The patients of dMCI have relatively focal dysfunction in executive domain with the tests of memory, language and visuospatial skills within normal limits. The patients with single domain dysexecutive MCI should meet the following criteria:

1. relatively focal executive dysfunction
2. Within reference range on tests of memory, language and visuospatial skills
3. normal general cognition
4. normal activities of daily living
5. not demented

The healthy volunteers

The healthy volunteers should be normal neuropsychological assessments as well as CDR=0 without significant neuropsychiatric disorder, right-handed, gender balanced and meet the following criteria:

1. Age and gender matched healthy subjects without significant neuropsychiatric disorder
2. Able to understand and provide signed informed consent

Exclusion Criteria:

The following exclusion criteria apply to all groups.

1. Cardiac pacemaker implantation.
2. Implantation of intracranial metal device.
3. Other major systemic disease, such as renal failure, heart failure, stroke, AMI/unstable angina, poor controlled diabetes mellitus, poor controlled hypertension.
4. Alcohol or drug abuse
5. Meet the criteria for dementia ( DSM-IV )
6. History of neurological disorder
7. Current psychiatrical illness
8. Head trauma with loss of consciousness greater than 10 minutes
9. Severe sensory deficit
10. Taking medication that affect cognition
11. Vascular lesion on MRI with Longstreth grade >=4
12. Structural abnormalities that could produce dementia, such as cortical infarction, tumor, or subdural hematoma
13. Treatments or concurrent illnesses other than Alzheimer disease that interfered with cognitive function.

Conversion Criteria

Patient with AD is not an enrolling group. The criteria as the MCI patients converted to is defined by NINCDS-ADRDA Criteria and CDR=0.5, 1 or 2. The diagnosis is based on the following:

1. CDR = 0.5, 1.0 or 2.0. For those of CDR 0.5, the diagnosis of MCI or AD depends on the judgment of the investigators on the level of clinical, ADL and neuropsychological impairment.
2. Probable AD defined by NINCDS/ADRDA criteria.
3. Caregiver/informant to accompany patient to all scheduled visits.
4. HAM-D rating scale score of 12 on the 17-item scale(19) or Cornell Scale for Depression in Dementia (CSDD) score<8(20).

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient will be recruited from the movement disorder clinics in ChangGung memorial hospital LinKou. The healthy control will be recruited from the local community in northem Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2011-01; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
differentiation of MCI using diffusion MRI | end of the first year
  The following will be measured in order to assess the diagnostic performance of diffusion MRI
  1. the sensitivity and specificity determined by Receiver operatic characteristic analysis
  2. the correlation between the neuropsychiatry batter and the measured diffusivity To determine the diagnostic sensitivity and specificity of MCI using diffusion MRI.
  With these two measurement, the outcome is to differentiate the subtypes of MCI

SECONDARY OUTCOMES:
Prognosis value of diffusion MRI | end of the third year
  The clinical deterioration will be determined by the difference in neuropsychiatry battery between the third year and the first year. The analysis will be made with and without the first year diffusion MRI. It will then be determined if the first year diffusion MRI can predict the decline in the third year. An optimal cutoff value will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Jiun-Jie Wang, PhD, Principal Investigator — ChangGung University
Locations (1):
- ChangGung Memorial Hospital, Linkou, Taoyuan District, Taiwan, Taiwan